CLINICAL TRIAL: NCT05563480
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQB2618 Injection Combined With Penpulimab in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: TQB2618 Injection Combined With Penpulimab Injection in the Treatment of Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-AK105-II-01
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-10

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Gemcitabine; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2618+Pempulimab+Chemotherapy (Experimental): Induction therapy: TQB2618 injection + Penpulimab injection + Gemcitabine hydrochloride injection + cisplatin injection; Maintenance treatment: TQB2618 injection +Penpulimab injection; 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 Injection, Pempulimab Injection, Cisplatin Injection, Gemcitabine Hydrochloride Injection
- Penpulimab + Chemotherapy (Active Comparator): Induction therapy: Penpulimab injection + Gemcitabine hydrochloride injection + cisplatin injection; Maintenance treatment: Penpulimab injection; 21 days as a treatment cycle.
  Interventions: Drug: Penpulimab injection, Cisplatin Injection, Gemcitabine Hydrochloride Injection
- TQB2618+Pempulimab (Experimental): TQB2618 injection combined with Penpulimab injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection; Penpulimab injection

INTERVENTIONS:
Drug: TQB2618 Injection, Pempulimab Injection, Cisplatin Injection, Gemcitabine Hydrochloride Injection — TQB2618 injection: Anti-TIM-3 monoclonal antibody; Penpulimab injection: Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1)
  Arms: TQB2618+Pempulimab+Chemotherapy
Drug: Penpulimab injection, Cisplatin Injection, Gemcitabine Hydrochloride Injection — Penpulimab injection: Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1)
  Arms: Penpulimab + Chemotherapy
Drug: TQB2618 injection; Penpulimab injection — TQB2618 injection: Anti-TIM-3 monoclonal antibody; Penpulimab injection: Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1)
  Arms: TQB2618+Pempulimab

SUMMARY:
This is a phase II clinical trial to evaluate the efficacy and safety of TQB2618 injection combined with Penpulimab in patients with recurrent/metastatic nasopharyngeal carcinoma.

This study is divided into two parts. The first part includes the safe introduction phase and the expansion phase. The second part is a randomized controlled study design, which is divided into two groups. The two parts of research are carried out at the same time

DETAILED DESCRIPTION:
This study is divided into two parts:

The first part includes the safe introduction phase and the expansion phase. All the patients with advanced nasopharyngeal carcinoma who failed to be treated with platinum chemotherapy and immunocheckpoint inhibitors (anti-PD-1 monoclonal antibody/anti-PD-L1 monoclonal antibody, etc.) were enrolled. The treatment scheme is TQB2618 + Penpulimab Injection. During the safe introduction period, we explored whether the two dose groups (1200mg/1500mg) were safe and tolerable when TQB2618 was combined with Penpulimab Injection. If the two dose groups are tolerable, 18~24 patients in the second phase of the extended study were randomized to receive TQB2618 in two dose groups (1200mg/1500mg)+Penpulimab Injection (200mg) at a ratio of 1:1. If high dose (1500mg) of TQB2618 is not tolerated, all patients will receive TQB2618 (1200mg)+Penpulimab Injection (200mg).

The second part is a randomized controlled study design, which is divided into two groups. All the newly treated patients with advanced nasopharyngeal carcinoma who have not received systematic treatment in the past received TQB2618+Penpulimab Injection+GP chemotherapy and paianzulimab+GP chemotherapy respectively. The dose of TQB2618 was 1200mg.

The two parts of research are carried out at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed nasopharyngeal carcinoma, stage IVb as defined by the AJCC TNM staging system for nasopharyngeal carcinoma, 8th edition in 2017 or subjects with recurrent nasopharyngeal carcinoma who were not suitable for local therapy (For neoadjuvant/adjuvant therapy and radical concurrent chemoradiotherapy, if the disease progresses during treatment or within 6 months after the treatment completion, it should be counted as a failure of first-line treatment of the original plan, and if it exceeds 6 months, it cannot be counted as first-line treatment failure. Alterations of treatment regimen due to drug intolerance are not defined as treatment failure).
* The first part of enrolled patients shall also meet the following requirements:

  1. At least received first-line treatment for recurrent/metastatic lesions, and the last anti-tumor treatment before enrollment had evidence of imaging progress in line with RECIST 1.1 standard;
  2. At least have received platinum containing chemotherapy and immunocheckpoint inhibitors (anti-PD-1 monoclonal antibody/anti-PD-L1 monoclonal antibody, etc.) in the past and failed treatment, and there is evidence of imaging progress that meets the RECIST 1.1 standard. Platinum containing chemotherapy and immunotherapy can be used during palliative treatment for recurrent/metastatic lesions, or during radical treatment for locally advanced diseases.
  3. Immunotherapy for recurrent/metastatic lesions shall not exceed 2 lines (For neoadjuvant/adjuvant therapy and radical concurrent chemoradiotherapy, if the disease progresses during treatment or within 6 months after the treatment completion, it should be counted as a failure of first-line treatment of the original plan, and if it exceeds 6 months, it cannot be counted as first-line treatment. Failure. Alterations of treatment regimen due to drug intolerance do not defined as treatment failure
  4. For the latest immunotherapy before enrollment, if it is aimed at recurrence/metastasis, the best efficacy is at least SD (≥ 6 weeks) or confirmed PR or immunotherapy duration ≥ 12 weeks.
* The second part of the enrolled patients also need to meet the following requirements:

  1. Have not received systemic antitumor therapy for recurrent/metastatic nasopharyngeal carcinoma before;
  2. No previous treatment with immune checkpoint inhibitors (anti PD-1 monoclonal antibody/anti PD-L1 monoclonal antibody, etc.). Those who have used no more than one immune checkpoint inhibitor (limited to CTLA-4/PD-1/PD-L1 monoclonal antibody, not including bispecific antibody, not including Penpulimab injection) in the stage of locally advanced radical treatment can be included if they meet the following criteria:

     1. If used in the induction phase (with or without other drugs), the best effect in the induction phase is at least PR;
     2. If used during radical radiochemotherapy/radiotherapy or subsequent maintenance stage, there is no progress during treatment and within one year after stopping treatment
* At least one measurable lesion confirmed according to RECIST 1.1 criteria;
* The function of main organs are well and meet the following standards:

  1. Routine Blood routine examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before the examination):

     1. Hemoglobin (HGB) ≥90 g/L;
     2. Absolute value of neutrophil (NEUT) ≥1.5×109/L;
     3. Platelets count (PLT) ≥ 100×109/L.
  2. The biochemical examination shall meet the following standards:

     1. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN) (Patients with Gilbert syndrome ≤ 3 × ULN);
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. If it is accompanied by liver metastasis, ALT and AST ≤ 5 × ULN;
     3. Serum creatinine (CR) ≤ 1.5 × ULN or Creatinine clearance (CCR) ≥ 60 ml/min;
  3. Blood coagulation function or thyroid function test should meet the following standards: Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulant therapy);
  4. Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, it can be selected.
  5. Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.
* Female subjects of reproductive age should agree that they must conduct contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during and for 6 months after the study; Female subjects should have a negative serum/urine pregnancy test within 7 days prior to study enrollment and must be non-lactating; Male subjects should agree that they must conduct contraception during the study period and for 6 months after the study.

Exclusion Criteria:

* Combined diseases and medical history:

  1. Other malignant tumors have occurred or are currently suffering from other malignant tumors within 5 years before the first medication, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ and papillary thyroid carcinoma;
  2. Unresolved toxicities greater than CTC AE grade 1 due to any prior therapy, excluding alopecia, neurotoxic sequelae associated with prior platinum therapy;
  3. Received major surgical treatment, obvious traumatic injury (excluding needle biopsy, endoscopic biopsy, etc.) within 28 days before the first drug;
  4. Arterial/venous thrombotic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months before the first drug;
  5. Active pulmonary tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or active pneumonia with clinical symptoms;
* Cancer-related symptoms and treatment:

  1. Received NMPA-approved Chinese patent medicines with anti-tumor indications in the drug insert within 2 weeks prior to the first administration;
  2. Received surgery, chemotherapy, radiotherapy or other anti-cancer therapy within 3 weeks before the start of study treatment (the washout period is calculated from the end of the last treatment); those who have received local radiotherapy in the past can be enrolled if they meet the following conditions: radiotherapy The end of the study treatment is more than 3 weeks (more than 2 weeks for brain radiotherapy); and the target lesions selected in this study are not in the radiotherapy area; Or the target lesion is located in the radiotherapy area, but the progress has been confirmed.
  3. Previous treatment with anti-TIM-3 antibodies;
  4. The nasopharyngeal lesions recurred after radiotherapy and received Re-radiotherapy;
  5. maging (CT or MRI) shows that the tumor has invaded around important blood vessels, and it is judged by the investigator that the tumor is very likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study;
  6. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
  7. Known uncontrolled or symptomatic active central nervous system (CNS) metastases presenting with clinical symptoms, cerebral edema, spinal cord compression, cancerous meningitis, leptomeningeal disease, and/or progressive growth. Patients with a history of CNS metastases or spinal cord compression were eligible if they were clearly treated and clinically stable after 4 weeks of discontinuation of anticonvulsants, steroids, or dehydrating agents prior to the first dose of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 3 weeks
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.
Objective Response Rate | Up to 60 weeks
  It is generally defined as complete response plus partial response.
Progression-free Survival | Up to 60 weeks
  The period between the beginning of treatment and the observation of disease progression or death from any cause in a patient with a tumor disease.

SECONDARY OUTCOMES:
Overall Survival | Baseline up to 100 weeks
  From drug use to the time of death from any cause.
Duration Of Response | 24 weeks
  It is the efficacy evaluation index of tumor response, which refers to the time from the first evaluation of tumor as complete response (CR) or partial response (PR) to the first evaluation of disease progression (PD) or death from any cause.
Disease Control Rate | Baseline up to 96 weeks
  It is the proportion of patients whose tumors have shrunk or stabilized for a certain amount of time and includes complete response (CR), partial response (PR), and stable (SD) cases.
Adverse Events | Baseline up to 100 weeks
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug.
Serious Adverse Event | Baseline up to 100 weeks
  It refers to adverse medical events such as death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization, and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital Sun Yat sen University, Zhuhai, Guangdong
  - Union Hospital Tongji Medical College, Huazhong University Of Science And Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No